CLINICAL TRIAL: NCT01552759
Title: Appetite Hormones in Binge Eating Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Obesity and Nutrition Research Center (Other)
Collaborators: St. Luke's-Roosevelt Hospital Center (Other); Columbia University (Other)
Responsible Party: Principal Investigator, Dr. Allan Geliebter, Principal Investigator, New York Obesity and Nutrition Research Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-163
Record Dates: First submitted 2012-03-09; First posted 2012-03-13 (Estimated); Last update posted 2013-03-11 (Estimated); Status verified 2013-03

CONDITIONS: Binge Eating Disorder
Keywords: Appetite Hormones; Binge Eating Disorder; Obesity; Cortisol; Stress
MeSH Terms: conditions — Binge-Eating Disorder; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Obese subjects with BED (Experimental): Subjects who meet the BMI requirement for obesity (>30 kg/m^2) and the DSM requirements for binge eating disorder based on responses to validated questionnaires.
  Subjects will undergo the postprandial responses, cold pressor test and ad libitum test meal.
  Interventions: Procedure: Postprandial responses; Behavioral: Cold pressor test; Behavioral: Test meal
- Obese without BED (Experimental): Subjects who meet the BMI requirement for obesity (>30 kg/m^2) but who do not meet the DSM requirements for binge eating disorder based on responses to validated questionnaires.
  Subjects will undergo the postprandial responses, cold pressor test and ad libitum test meal.
  Interventions: Procedure: Postprandial responses; Behavioral: Cold pressor test; Behavioral: Test meal
- Normal-weight without BED (Experimental): Subjects with BMI 20-25 kg/m^2 who do not meet the DSM requirements for binge eating disorder based on responses to validated questionnaires.
  Subjects will undergo the postprandial responses, cold pressor test and ad libitum test meal.
  Interventions: Procedure: Postprandial responses; Behavioral: Cold pressor test; Behavioral: Test meal

INTERVENTIONS:
Procedure: Postprandial responses — Subjects ingest a fixed meal, with blood draws to measure appetite hormone levels taken before and after the meal.
  Other Names: Liquid meal replacement is Boost (Nestle Nutrition).
Behavioral: Cold pressor test — Subjects then undergo the Socially-Evaluated Cold Pressor Test, with blood draws to measure appetite hormone levels taken before and after the test.
Behavioral: Test meal — Subjects are presented with an ad libitum buffet meal.

SUMMARY:
This study investigates the hormones that the body produces in response to food intake and in response to stress, and the way that stress influences food intake. In particular, it compares the hormone levels and food intake of people with and without binge eating disorder. In order to find out how these appetite- and stress-related hormones are linked to brain activity, the study also includes an fMRI scan, a non-invasive procedure that looks at which regions of the brain are most active during a food-related scenario.

DETAILED DESCRIPTION:
The objectives are to study appetite-related hormones regulating food intake under normal conditions and following a stressor in the morning and evening (when most binge episodes occur), to help reveal biological mechanisms in BED. We plan to enroll: 32 obese Ss with BED (16m, 16f), 32 obese Ss without BED (16m, 16f) and 32 normal-weight Ss without BED (16m, 16f). Height, weight, waist circumference, and body fat will be assessed during a first appointment. On two different days separated by at least a week, Ss will ingest a fixed liquid meal once in the morning and once in the evening. Appetite ratings and collections of blood and saliva to measure hormones will continue for 2 hours after the fixed meal. This will be followed on each day by a laboratory stress protocol (Socially Evaluated Cold Pressor Test; SECPT), and then consumption of an ad libitum meal 30 minutes later. On one day during the protocol, the participant will collect saliva using a swab immediately after waking and again at 08.00. In order to capture more naturalistic eating episodes, all Ss will additionally record food intake, rate appetite, and measure salivary cortisol before and after one evening meal, and one after-dinner snack (or after-dinner binge for BED Ss). On two additional days, we will use fMRI to assess brain activation in response to high-palatability food (HPF) relative to low-palatability food (LPF) or non-food (NF) visual cues following the SECPT and a control condition using warm water. On each day, following the fMRI scan, an ad libitum meal will be consumed.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 20-25 or 30-50
* stable weight(± 4%) for at least 3 mo
* premenopausal and have regular menstrual cycles (28 d ± 5), not be pregnant or lactating, and not be within 1 y of childbirth
* must like pizza and be willing to consume it during the ad libitum meal

Exclusion Criteria:

* significant medical or psychiatric conditions
* current and past 3-mo use of certain prescribed medications, especially those that could affect body weight, such as antidepressants and stimulants as well as smoking, or excess alcohol (> 3 drinks/d)
* vigorously exercise for more than 6 h/wk
* left-handed, with known claustrophobia for a scanner enclosure, or have metal implants, non-removable metallic dental retainers, pacemakers, or permanent eyeliner or large tattoos that contain metallic pigment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2007-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Appetite-related Hormones and Appetite Ratings in Relation to Fixed Meal and Cold Pressor Test | Assessed at systematic intervals (-15, 0, 10, 30, 60, 90, 120 min) before and after the morning fixed meal at 10.00 and the evening fixed meal at 17.00
  Blood and saliva concentrations of hormones influencing appetite will be measured at systematic intervals (-15, 0, 10, 30, 60, 90, 120 min) before and after the morning fixed meal at 10.00 and the evening fixed meal at 17.00. Appetite will additionally be rated at each assessment point. This will be followed by a cold pressor test, and then 30 min later by an ad libitum meal 30 min later, with blood and saliva measurements taken before and after completion of the meal.

SECONDARY OUTCOMES:
Cortisol Awakening response | Assessed on one weekday morning during the 3-week participation period
  On one weekday morning during the 3-week participation period, participants will take one saliva measurement on awakening and at 08.00 while still fasting. Awakening and 08.00 cortisol levels are expected to be higher in BED compared with nonBED Ss, and in obese nonBED compared with normal-weight nonBED Ss.
Psychological Scales | During one initial consultation and on two subsequent visits at least 1 week apart
  Various questionnaires will be administered to test relationships between outcomes (e.g., intake, hormone levels), and psychological constructs including depression, perceived stress, external and emotional eating and restraint, binge-eating behavior, and night eating. Outcomes will be correlated with scale scores, and scores will be compared between groups. Among other relationships, we anticipate positive correlations between binge eating score, ad libitum intake and ghrelin SECPT response. Psychological scores will be entered as covariates as appropriate.
Body Weight, Body Composition and Gender | During one initial consultation and on two subsequent visits at least 1 week apart
  Measurements will include height, weight, waist circumference, total body fat from BIA, and cross-sectional abdominal MRI to estimate central, visceral, and subcutaneous fat. Each adiposity index will be correlated with outcomes and compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Allan Geliebter, PhD, Principal Investigator — New York Obesity and Nutrition Research Center
Locations (1):
- St. Luke's Hospital, New York, New York, United States

REFERENCES:
- [Background] de Zwaan M, Mitchell JE, Raymond NC, Spitzer RL. Binge eating disorder: clinical features and treatment of a new diagnosis. Harv Rev Psychiatry. 1994 Mar-Apr;1(6):310-25. doi: 10.3109/10673229409017098. PMID 9384866
- [Background] Hellstrom PM, Geliebter A, Naslund E, Schmidt PT, Yahav EK, Hashim SA, Yeomans MR. Peripheral and central signals in the control of eating in normal, obese and binge-eating human subjects. Br J Nutr. 2004 Aug;92 Suppl 1:S47-57. doi: 10.1079/bjn20041142. PMID 15384323
- [Background] Cowley MA, Smith RG, Diano S, Tschop M, Pronchuk N, Grove KL, Strasburger CJ, Bidlingmaier M, Esterman M, Heiman ML, Garcia-Segura LM, Nillni EA, Mendez P, Low MJ, Sotonyi P, Friedman JM, Liu H, Pinto S, Colmers WF, Cone RD, Horvath TL. The distribution and mechanism of action of ghrelin in the CNS demonstrates a novel hypothalamic circuit regulating energy homeostasis. Neuron. 2003 Feb 20;37(4):649-61. doi: 10.1016/s0896-6273(03)00063-1. PMID 12597862
- [Background] Batterham RL, Cohen MA, Ellis SM, Le Roux CW, Withers DJ, Frost GS, Ghatei MA, Bloom SR. Inhibition of food intake in obese subjects by peptide YY3-36. N Engl J Med. 2003 Sep 4;349(10):941-8. doi: 10.1056/NEJMoa030204. PMID 12954742
- [Background] English PJ, Ghatei MA, Malik IA, Bloom SR, Wilding JP. Food fails to suppress ghrelin levels in obese humans. J Clin Endocrinol Metab. 2002 Jun;87(6):2984. doi: 10.1210/jcem.87.6.8738. PMID 12050284
- [Background] Monteleone P, Martiadis V, Rigamonti AE, Fabrazzo M, Giordani C, Muller EE, Maj M. Investigation of peptide YY and ghrelin responses to a test meal in bulimia nervosa. Biol Psychiatry. 2005 Apr 15;57(8):926-31. doi: 10.1016/j.biopsych.2005.01.004. PMID 15820714
- [Background] Monteleone P, Martiadis V, Fabrazzo M, Serritella C, Maj M. Ghrelin and leptin responses to food ingestion in bulimia nervosa: implications for binge-eating and compensatory behaviours. Psychol Med. 2003 Nov;33(8):1387-94. doi: 10.1017/s0033291703008316. PMID 14672247
- [Background] Geliebter A, Yahav EK, Gluck ME, Hashim SA. Gastric capacity, test meal intake, and appetitive hormones in binge eating disorder. Physiol Behav. 2004 Jul;81(5):735-40. doi: 10.1016/j.physbeh.2004.04.014. PMID 15234178
- [Background] Geliebter A, Gluck ME, Hashim SA. Plasma ghrelin concentrations are lower in binge-eating disorder. J Nutr. 2005 May;135(5):1326-30. doi: 10.1093/jn/135.5.1326. PMID 15867334
- [Background] Raymond NC, Neumeyer B, Warren CS, Lee SS, Peterson CB. Energy intake patterns in obese women with binge eating disorder. Obes Res. 2003 Jul;11(7):869-79. doi: 10.1038/oby.2003.120. PMID 12855757
- [Background] Walsh BT, Boudreau G. Laboratory studies of binge eating disorder. Int J Eat Disord. 2003;34 Suppl:S30-8. doi: 10.1002/eat.10203. PMID 12900984
- [Background] Anderson DA, Williamson DA, Johnson WG, Grieve CO. Validity of test meals for determining binge eating. Eat Behav. 2001 Summer;2(2):105-12. doi: 10.1016/s1471-0153(01)00022-8. PMID 15001040
- [Background] Geliebter A, Melton PM, McCray RS, Gallagher DR, Gage D, Hashim SA. Gastric capacity, gastric emptying, and test-meal intake in normal and bulimic women. Am J Clin Nutr. 1992 Oct;56(4):656-61. doi: 10.1093/ajcn/56.4.656. PMID 1414964
- [Background] Geliebter A, Hassid G, Hashim SA. Test meal intake in obese binge eaters in relation to mood and gender. Int J Eat Disord. 2001 May;29(4):488-94. doi: 10.1002/eat.1047. PMID 11285588
- [Background] Tataranni PA, Larson DE, Snitker S, Young JB, Flatt JP, Ravussin E. Effects of glucocorticoids on energy metabolism and food intake in humans. Am J Physiol. 1996 Aug;271(2 Pt 1):E317-25. doi: 10.1152/ajpendo.1996.271.2.E317. PMID 8770026
- [Background] Castonguay TW. Glucocorticoids as modulators in the control of feeding. Brain Res Bull. 1991 Sep-Oct;27(3-4):423-8. doi: 10.1016/0361-9230(91)90136-8. PMID 1959040
- [Background] Epel E, Lapidus R, McEwen B, Brownell K. Stress may add bite to appetite in women: a laboratory study of stress-induced cortisol and eating behavior. Psychoneuroendocrinology. 2001 Jan;26(1):37-49. doi: 10.1016/s0306-4530(00)00035-4. PMID 11070333
- [Background] Koo-Loeb JH, Costello N, Light KC, Girdler SS. Women with eating disorder tendencies display altered cardiovascular, neuroendocrine, and psychosocial profiles. Psychosom Med. 2000 Jul-Aug;62(4):539-48. doi: 10.1097/00006842-200007000-00013. PMID 10949100
- [Background] Kelly CB, Cooper SJ. Plasma norepinephrine response to a cold pressor test in subtypes of depressive illness. Psychiatry Res. 1998 Oct 19;81(1):39-50. doi: 10.1016/s0165-1781(98)00086-9. PMID 9829649
- [Background] Gluck ME, Geliebter A, Hung J, Yahav E. Cortisol, hunger, and desire to binge eat following a cold stress test in obese women with binge eating disorder. Psychosom Med. 2004 Nov-Dec;66(6):876-81. doi: 10.1097/01.psy.0000143637.63508.47. PMID 15564352
- [Background] Yanovski SZ. Binge eating disorder: current knowledge and future directions. Obes Res. 1993 Jul;1(4):306-24. doi: 10.1002/j.1550-8528.1993.tb00626.x. PMID 16350580
- [Background] Geliebter A, Ladell T, Logan M, Schneider T, Sharafi M, Hirsch J. Responsivity to food stimuli in obese and lean binge eaters using functional MRI. Appetite. 2006 Jan;46(1):31-5. doi: 10.1016/j.appet.2005.09.002. Epub 2005 Dec 20. PMID 16364498
- See also: New York Obesity and Nutrition Research Center — http://www.nyorc.org/